CLINICAL TRIAL: NCT02625883
Title: Out-of-Hospital Resuscitation in an Urban Setting in Switzerland - an Outcome Study and Cost Effectiveness Analysis
Brief Title: Out-of-Hospital Resuscitation in Winterthur - an Outcome Study
Status: Completed | Type: Observational
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Other Study IDs: Resuscitation in Winterthur
Record Dates: First submitted 2015-12-07; First posted 2015-12-09 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Resuscitation
Keywords: Resuscitation, quality of life
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survivors: Patients with out-of-Hospital resuscitation and return of spontaneous circulation. Structured interview for quality of life (questionnaire) one year after resuscitation.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Interview by validated Quality-of-life-questionnaire
  Other Names: patient interviews

SUMMARY:
The investigators will retrospectively examine all patients with out-of-hospital resuscitation by the emergency medical Team (EMT) from the Kantonsspital Winterthur in the year 2013 with a two year follow-up and a structured interview about Quality of life. Furthermore, the costs generated by the local health system are analysed.

DETAILED DESCRIPTION:
The Primary objective of this study is to evaluate the Quality of out-of-Hospital resuscitation by the ambulance Service from the Kantonsspital Winterthur including a 2-year follow-up of the survivors. In this follow-up we evaluate the Quality of life by a validated questionnaire.

The following endpoints will be retrospectively analysed:

time-to-Response Interval; Initial cardiac rhythm; medications given; number of Defibrillations; return of spontaneous circulation, Overall costs for the local health System

Furthermore length of hospital-stay, survival until Hospital discharge, one-year survival, Quality of life two years after resuscitation and total costs will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with out-of-hospital resuscitation in Winterthur in the year 2013 and treatment by the emergency medical team from the Kantonsspital Winterthur
* Written informed consent of patients for structured interview

Exclusion Criteria:

* Patients with resuscitation but death on Scene
* no written informed consent from patients for structured interview

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that were resuscitated out-of-hospital in the year 2013 by the emergency medical team from the Kantonsspital Winterthur.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Survival after prehospital cardiac Arrest until discharge of Hospital and a one-year follow-up | 1 year

SECONDARY OUTCOMES:
Evaluation of direct costs of local health care system | 1 year
Quality of life one year after resuscitation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ganter, director, Principal Investigator — sponsor and principal investigator

REFERENCES:
- [Derived] Ruch R, Stoessel L, Stein P, Ganter MT, Button DA. Outcome, quality of life and direct costs after out-of-hospital cardiac arrest in an urban region of Switzerland. Scand J Trauma Resusc Emerg Med. 2019 Nov 27;27(1):106. doi: 10.1186/s13049-019-0682-7. PMID 31771619